CLINICAL TRIAL: NCT02092298
Title: A Phase II Study of Laparoscopic Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) for Gastric Carcinomatosis or Positive Cytology
Brief Title: Laparoscopic Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) for Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0989; NCI-2014-01105 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal cancer; Hyperthermic Intraperitoneal Chemoperfusion; HIPEC; Gastric carcinomatosis; Gastroesophageal cancer; Mitomycin C; Mitomycin; Cisplatin; Platinol-AQ; Platinol; CDDP; Sodium Thiosulfate; Tinver
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Mitomycin; Cisplatin; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hyperthermic Intraperitoneal Chemotherapy (HIPEC) (Experimental): Laparoscopic HIPEC consists of Mitomycin C 30 mg and Cisplatin 200 mg for 60 minutes, performed 2-8 weeks after completion of systemic chemotherapy. Loading dose Sodium Thiosulfate 7.5 gm/M2 infused prior to addition of Cisplatin to the peritoneal perfusion circuit. Then a maintenance infusion of Sodium Thiosulfate 25.56 gm/M2 delivered by infusion pump over 12 hours.
  Interventions: Drug: Mitomycin C; Drug: Cisplatin; Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Mitomycin C — Mitomycin C 30 mg delivered laparoscopically for 60 minutes.
  Other Names: Mitomycin
Drug: Cisplatin — Cisplatin 200 mg delivered laparoscopically 60 minutes, 2-8 weeks after completion of systemic chemotherapy.
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Sodium Thiosulfate — Loading dose of 7.5 gm/M2 of Sodium Thiosulfate infused prior to addition of Cisplatin to the peritoneal perfusion circuit. Then a maintenance infusion of Sodium Thiosulfate 25.56 gm/M2 delivered by continuous infusion pump over 12 hours.
  Other Names: Tinver

SUMMARY:
The goal of this clinical research study is to learn if hyperthermic intraperitoneal chemotherapy (HIPEC) will help to control the disease in patients with Stage 4 stomach or gastroesophageal cancer. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
HIPEC Treatment:

If you are found to be eligible to take part in this study, on the day of HIPEC treatment, you will receive heated mitomycin-C and cisplatin as a liquid that is injected through 3 to 4 small incisions in your abdomen for about 1 hour. This will be done as a surgical procedure, and you will be under general anesthesia. The chemotherapy will then be flushed out of your abdomen and collected, and the treatment area inside your abdomen will be washed. Also during the HIPEC procedure, fluid will be collected and checked for cancer cells. As is standard of care, any lesions that are found during treatment may also be biopsied at this time, if the study doctor thinks it is necessary. You may receive up to 5 HIPEC treatments on this study.

You will also receive sodium thiosulfate by vein over about 20 minutes to protect the kidneys.

You will remain in the hospital for 3-7 days after treatment.

While you are in the hospital after surgery:

* Blood (about 2-3 tablespoons) may be drawn for routine tests, if the study doctor thinks it is necessary.

Study Visits:

One (1) time between Weeks 2-6:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.

Gastrectomy Surgery:

If your doctor thinks it is needed, you will have a standard of care surgery. You will receive a separate consent form which explains the surgery and its risks.

On or before 8 weeks after your surgery:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.

Follow-Up Visits:

You will have routine clinic visits every 6 months from the date of your last surgery. You will be asked about any other cancer treatments you may be receiving. If you stopped the study early, the study doctor may ask you to return to the office for extra CT scans, PET scan, or MRIs during the follow-up period.

You will have a CT scan, PET scan, or MRI of your chest, abdomen, and pelvis every 6 months for 5 years after surgery to check the status of the disease.

Length of Study Participation:

You will be on study for about 5 years after your last surgery. You will be taken off study early if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

This is an investigational study. The chemotherapy and surgery are standard treatment for stomach and gastroesophageal cancer. It is investigational to give the chemotherapy by HIPEC.

Up to 30 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above. There will be no upper age restriction.
2. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
3. Cytologic or histologic proof of adenocarcinoma of the stomach or gastroesophageal junction.
4. Adequate renal, and bone marrow function: a. Leukocytes >/= 3,000/microL; b. Absolute neutrophil count >/= 1,500/microL; c. Platelets >/= 100,000/Ul; d. Serum creatinine </= 1.5 mg/dL.
5. Hepatic function: AST (SGOT)/ALT (SGPT) </= 5 X institutional (Upper Limit of Normal) ULN.
6. Distant Metastatic Disease limited to peritoneum and radiologically occult (not visualized on preoperative imaging to include [Computerized Tomography] CT scan, Ultrasound, [Magnetic Resonance Imaging] MRI, PET/CT): a. Positive peritoneal cytology; b. Carcinomatosis on diagnostic laparoscopy or laparotomy.
7. Completion of preoperative systemic chemotherapy.

Exclusion Criteria:

1. Distant metastatic disease not limited to peritoneum: a. Solid organ metastases (liver, central nervous system, lung).
2. Any distant metastatic disease visualized on preoperative imaging: a. Solid organ metastases; b. Clear radiologic evidence of carcinomatosis.
3. Infections such as pneumonia or wound infections that would preclude protocol therapy.
4. Women with a positive urine or serum pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to refrain from breast feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence.
5. Subjects with unstable angina or New York Heart Association Grade II or greater congestive heart failure.
6. Subjects deemed unable to comply with study and/or follow-up procedures.
7. Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-05-08 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D. Badgwell, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Badgwell B, Blum M, Das P, Estrella J, Wang X, Fournier K, Royal R, Mansfield P, Ajani J. Lessons learned from a phase II clinical trial of laparoscopic HIPEC for gastric cancer. Surg Endosc. 2018 Jan;32(1):512. doi: 10.1007/s00464-017-5668-9. Epub 2017 Jun 22. PMID 28643069
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2014-July 2016. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: A total of 21 participants were consented, 2 participants were screen failures
Period: Overall Study
Arm/Group | Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 51 [35 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) After Hyperthermic Intraperitoneal Chemotherapy
Description: Primary objective of study is to assess overall survival (OS) in subjects with stage IV gastric cancer representing positive cytology or imaging occult carcinomatosis after laparoscopic hyperthermic intraperitoneal chemotherapy administration. Overall survival measured from time of laparoscopic HIPEC. Patterns of tumor recurrence and survival assessed by reviewing routine surveillance CT scans. Overall survival time estimated using the Kaplan-Meier method.
Time Frame: Between the second and sixth week after treatment, up to 5 years
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Number analyzed (Participants) | 19
Months | 30.2 (18.3)

2. Primary Outcome: Overall Survival (OS) From the First Laparoscopic HIPEC
Description: Primary objective of study is to assess overall survival (OS) in subjects with stage IV gastric cancer representing positive cytology or imaging occult carcinomatosis after the first laparoscopic HIPEC. Patterns of tumor recurrence and survival assessed by reviewing routine surveillance CT scans. Overall survival time estimated using the Kaplan-Meier method.
Time Frame: From the day of surgery, until the last day of follow up, until death, up to 5 years
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Number analyzed (Participants) | 19
Months | 20.3 (7.2)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious Adverse Events) for 30 days and All-Cause Mortality for 5 years
Arm/Group | Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
All-Cause Mortality (participants affected / at risk) | 18/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 4/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperthermic Intraperitoneal Chemotherapy (HIPEC) (N=19)
Arrythmia (Cardiac disorders) | 1
Kidney dysfunction (Renal and urinary disorders) | 1
Lung Injury (Respiratory, thoracic and mediastinal disorders) | 1
Blood Clot (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT02092298/Prot_SAP_000.pdf